CLINICAL TRIAL: NCT04192019
Title: Subcutaneous Dasiglucagon Use During Exercise In People With Type 1 Diabetes: Effects On Plasma Glucose And Exercise Metabolism
Brief Title: Micro Glucagon During Exercise in Type 1 Diabetes
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Prioritization of other projects
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: GLU-01
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: type 1 diabetes; glucagon; hypoglycemia; exercise; glycogen
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Motor Activity | interventions — dasiglucagon

STUDY DESIGN:
Intervention Model Description: Time to hypoglycaemia during 60 minutes of aerobic exercise in individuals with type 1 diabetes using mini and micro doses of Dasiglucagon compared to no Dasiglucagon
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Micro-dose glucagon (Experimental): 80 µg (micro-dose) subcutaneous Dasiglucagon 5 min before the start of exercise
  Interventions: Drug: Micro-glucagon
- Mini-dose glucagon (Experimental): 150 µg mini-dose of subcutaneous Dasiglucagon 5 min before exercise the start of exercise
  Interventions: Drug: Mini-glucagon
- No treatment (No Intervention): No treatment before the start of exercise

INTERVENTIONS:
Drug: Micro-glucagon — Administration of 80 µg (micro-dose) subcutaneous Dasiglucagon 5 min before the start of exercise
  Other Names: Dasiglucagon
  Arms: Micro-dose glucagon
Drug: Mini-glucagon — Administration of 150 µg (mini-dose) subcutaneous Dasiglucagon 5 min before the start of exercise
  Other Names: Dasiglucagon
  Arms: Mini-dose glucagon

SUMMARY:
This proof-of-principle study to assess effects of different doses (mini and micro) of subcutaneous glucagon analog Dasiglucagon (Zealand Pharma, Copenhagen, Denmark) on the change in blood glucose concentration during moderate-intensity exercise in people with T1D.

DETAILED DESCRIPTION:
People with type 1 diabetes (T1D) are recommended to engage in regular exercise for a variety of health and fitness reasons. However, moderate-intensity exercise is associated with an increased risk of hypoglycaemia in people with T1D. Current guidelines are to reduce insulin dose and/or increase carbohydrate consumption in the context of the exercise bout. However, despite the many advances in insulin formulations and delivery devices, hypoglycaemia remains a significant risk. Mini-dose glucagon taken before an exercise bout has been shown to be an effective non-caloric strategy to prevent exercise-induced hypoglycaemia. However, even the reduced doses (150-200 µg) used in previous studies might still be rather high translating into potential side-effects (i.e. hyperglycaemia, gastrointestinal symptoms, etc.). Lower doses (below 100 µg, micro-glucagon) may be sufficiently effective to counteract hypoglycaemia risk associated with exercise and associated with better tolerance. Moreover, there is little information on the effects of subcutaneous glucagon on glycogen stores and changes in exercise metabolism. Greater understanding of exercise-associated metabolism following mini- and micro-dose glucagon using techniques such as magnetic resonance spectroscopy (MRS), continuous glucose monitoring (CGM), stable isotope tracers, and indirect calorimetry may result in novel approaches to improve blood glucose management in people with T1D. Utilising these techniques may also further our understanding of the optimal glucagon dosing (timing and amount) during exercise to manage hypoglycaemia and reduce the risk of adverse events. Proof-of-principle study to assess effects of different doses (mini and micro) of subcutaneous glucagon analog Dasiglucagon (Zealand Pharma, Copenhagen, Denmark) on the change in blood glucose concentration during moderate-intensity exercise in people with T1D. Secondly, to investigate exercise-metabolism following Dasiglucagon injection using 3 tesla magnetic resonance spectroscopy (MRS) and indirect calorimetry. Third, to assess participant experience of Dasiglucagon during exercise and the incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* T1D for >1 year
* Male aged 18-45 years old
* HbA1c <8.0% (64 mmol/mol) based on analysis from the central laboratory unit of Bern University Hospital
* Regular physical activity (defined as meeting 150 min moderate-intensity exercise per week)
* Using either continuous subcutaneous insulin infusion or multiple daily injections
* Written informed consent

Exclusion Criteria:

* Physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the results as judged by the investigator
* Current treatment with drugs known to interfere with metabolism e.g. systemic corticosteroids, statins, SGLT2 inhibitors, GLP1 agonists
* Relevant diabetic complications as judged by the investigator
* Body mass index 30 kg/m2
* Uncontrolled hypertension (>180/100 mmHg)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Time to hypoglycaemia | 60 minutes
  Time (in minutes) to hypoglycaemia (plasma glucose <3.9mmol/l) during 60 minutes of aerobic exercise in individuals with type 1 diabetes using mini and micro doses of Dasiglucagon compared to no Dasiglucagon

SECONDARY OUTCOMES:
Change in glycaemia during exercise | 60 minutes
  Change in blood glucose concentration, calculated based on the participants' glucose at the start of exercise and the last value measured at the end of exercise. If the exercise is stopped early because of hypoglycaemia, the last exercise glucose value will be used for analysis
Glucose during exercise | 60 minutes
  Mean glucose concentration and area under the glucose curve during exercise
Glucagon during exercise | 60 minutes
  Mean glucagon concentration and area under the glucagon curve during exercise
Time in target | 24 hours
  Time in target glycaemic range (4-10 mmol/L) in the recovery period and overnight
Time in target during exercise | 60 minutes
  Time in target glycaemic range (4-10 mmol/L) during exercise
Hypoglycaemia | 24 hours
  Incidence of hypoglycaemia (≤3.9 mmol/L for 15 min or more) during the 24 hour post exercise recovery period
Glycogen content | 4 hours
  Change in skeletal muscle and hepatic glycogen following exercise
Any adverse events | 24 hours
  Adverse symptoms following glucagon/placebo use

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stettler, MD, Principal Investigator — Clinic Director

IPD SHARING:
Plan to Share IPD: No